CLINICAL TRIAL: NCT02351206
Title: Lumbar Intervertebral Disc Space Height in Disc Herniation and Degeneration Patients in Their Early 20s
Brief Title: Lumbar Disc Space Height in Young Disc Herniation and Degeneration Patients
Status: Completed | Type: Observational
Sponsor: Jaseng Hospital of Korean Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: JS-CT-2014-05
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Intervertebral Disc Displacement; Intervertebral Disc Degeneration; Low Back Pain
Keywords: X-Rays; Magnetic Resonance Imaging; Sensitivity and Specificity
MeSH Terms: conditions — Intervertebral Disc Displacement; Intervertebral Disc Degeneration; Low Back Pain; Hypersensitivity | interventions — X-Rays; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- The experimental group: Patients with intervertebral disc protrusion, extrusion, or migration at L4/5 randomly selected from a population pool of 665 patients with L-spine X-ray and L-spine MRIs taken within a week of the other test.
  Interventions: Radiation: x-ray, MRI
- The control group: Patients with normal or disc bulging readings at L4/5 randomly selected from a population pool of 665 patients with L-spine X-ray and L-spine MRIs taken within a week of the other test.
  Interventions: Radiation: x-ray, MRI

INTERVENTIONS:
Radiation: x-ray, MRI

SUMMARY:
As low back pain (LBP) imposes a heavy socioeconomic burden, early detection of pathologic intervertebral disc change in young adults holds high clinical relevance as a common structural cause of LBP. The investigators therefore assessed the feasibility of using X-ray disc space height measurements as a predictive evaluation method of lumbar disc herniation (LDH) and degeneration in LBP patients in their early 20s.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-25 years
* L-spine X-ray and L-spine MRIs taken within a week of the other test
* Native Korean ethnicity

Exclusion Criteria:

* Scoliosis with a Cobb's angle of ≥20°
* Significant vertebral deformity of any etiology (e.g. spondylolisthesis, fracture, spondylitis, neoplasm)
* Previous spinal surgery

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients visiting Jaseng hospital of Korean Medicine, a spine specializing Korean medicine hospital designated by the Korean ministry of health and welfare, from January, 2010 to October 2014
Sampling Method: Probability Sample
Enrollment: 389 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The distance between the 2 midpoints of the inferior and superior borders of the vertebral bodies surrounding the L4/5 intervertebral disc space divided by the AP diameter of the inferior border of the L4 vertebral body | Baseline